CLINICAL TRIAL: NCT06476366
Title: Comparison of Efficacy of Methotrexate and Azathioprine in Patients With Chronic Actinic Dermatitis
Brief Title: Comparison of Efficacy of Methotrexate and Azathioprine in Patients With Chronic Actinic Dermatitis: A Randomized Controlled Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ahsan Tameez-ud-din, Registrar Dermatology, Pak Emirates Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DERM9512866
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Chronic Actinic Dermatitis
MeSH Terms: conditions — Photosensitivity Disorders | interventions — Azathioprine; Methotrexate

STUDY DESIGN:
Intervention Model Description: Two arms of the study will be as follows:
  Group A: Methotrexate 10mg/week Group B: Azathioprine 0.3mg/kg daily
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate arm (Active Comparator): After the enrollment of patients and taking consent, participants will be divided in two treatment groups via lottery method. Group A will be administered oral methotrexate 10mg/week after a test dose. Starting dose will be 2.5mg/week and dose will be escalated by 2.5mg/week till the final dose of 10mg/week
  Interventions: Drug: Methotrexate
- Azathioprine (Active Comparator): group B will be administered tablet azathioprine at a dose of 0.3mg/kg daily after TPMT testing. Both group of patients will be advised regarding strict sun protection measures (sunblock, hats, sunglasses etc.). The baseline investigations for both groups will include complete blood picture (CBC), liver function tests (LFTs), renal function tests (RFTs), electrocardiogram, chest X-ray and urine analysis while thiopurine methyltransferase (TPMT) levels will be assessed specifically for group B patients. The patients will be followed up at week 4, 12 and 24. CBC, RFTs and LFTs will be done at each follow-up and EASI score will be calculated,
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Azathioprine — azathioprine will be started at 0.3mg/kg orally daily. Anticipated response is after atleast 1 month so testing will be done thereafter ( after checking TPMT levels)
  Arms: Azathioprine
Drug: Methotrexate — Methotrexate will be started at 5mg/week and dose escalated by 2.5mg weekly to ultimately 10mg/week. Tablet Folic acid 0.5mg will be given orally daily, skipping the day of methotrexate
  Arms: Methotrexate arm

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of AZT and MTX in patients with Chronic Actinic Dermatitis (CAD). These drugs have been used successfully as steroid-sparing alternatives in a variety of related dermatoses and this trial may help in paving the path towards the ubiquitous use of these cost-effective and relatively safer drugs in CAD patients of our population. The researchers will try to answer the following questions:

1. Is methotrexate safe and efficacious in treating CAD?
2. Is there a difference in efficacy of methotrexate and azathioprine in the treatment of this disease?

After the enrollment of patients and taking consent, participants will be divided in two treatment groups via lottery method. Group A will be administered oral methotrexate 10mg/week after a test dose while group B will be administered tablet azathioprine at a dose of 0.3mg/kg daily after. Both group of patients will be advised regarding strict sun protection measures (sunblock, hats, sunglasses etc.). The baseline investigations for both groups will include complete blood picture (CBC), liver function tests (LFTs), renal function tests (RFTs), electrocardiogram, chest X-ray and urine analysis while thiopurine methyltransferase (TPMT) levels will be assessed specifically for group B patients. The patients will be followed up at week 4, 12 and 24. CBC, RFTs and LFTs will be done at each follow-up and Eczema Area and Severity Index (EASI) score will be calculated, Investigator global assesment (IGA) score will also be calculated .

DETAILED DESCRIPTION:
Weekly complete blood picture (CBC) will be done until the last dose escalation for group B patients. Both group of patients will be advised regarding strict sun protection measures (sunblock, hats, sunglasses). The baseline investigations for both groups included CBC, liver function tests (LFTs), renal function tests (RFTs), electrocardiogram, chest X-ray and urine analysis while TPMT levels will be assessed specifically for group B patients. The patients will be followed up at week 4, 12 and 24. CBC, RFTs and LFTs will be done at each follow-up. EASI score will be calculated at baseline and at subsequently at each follow-up visit.

A comparison from the EASI score from the last visit will be made at each follow-up to assess whether any patient achieved the primary outcome of EASI-50 (50% improvement in EASI score from baseline). Investigator global assessment (IGA) score will be used as a secondary outcome measure. It is a subjective measure of disease severity which is assessed by the physician on patient's every visit. It ranges from 0 to 4 (0-clear, 1-almost clear, 2-mild, 3-moderate, 4-severe). An IGA score of 0-2 will be considered as the outcome measure. Patients will be also asked for any specific side-effects of the treatment at every follow-up. The data including the demographic profile of the participants will be recorded on a printed form. The data will be kept under lock and key and will be available only to the treating physician and the research team.

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed as well as patients with an established diagnosis of CAD presenting to the outpatient department or the emergency department of PEMH or CMH will be included in the study.

Exclusion Criteria:

* Patients with coexisting conditions requiring immunosuppressants will be excluded from the study. Patients with dementia or any other neuropsychiatric disorder will also be excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahsan Tameez-ud-din, Principal Investigator — Pak Emirates Military Hospital
Locations (1):
- Pak Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
No plan to share the data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 patients recruited in each arm after informed consent as detailed in the attached document
Pre-assignment Details: Group A was administered oral methotrexate 10mg/week after a test dose while group B was administered tablet azathioprine at a dose of 0.3mg/kg daily after testing for TPMT levels. Both group of patients were advised regarding strict sun protection measures (sunblock, hats, sunglasses). The baseline investigations for both groups included complete blood picture (CBC), liver function tests (LFTs), renal function tests (RFTs), electrocardiogram, chest X-ray and urine analysis
Groups:
- Methotrexate Arm: After the enrollment of patients and taking consent, participants will be divided in two treatment groups via lottery method. Group A will be administered oral methotrexate 10mg/week after a test dose
- Azathioprine: group B will be administered tablet azathioprine at a dose of 0.3mg/kg daily after. Both group of patients will be advised regarding strict sun protection measures (sunblock, hats, sunglasses etc.). The baseline investigations for both groups will include complete blood picture (CBC), liver function tests (LFTs), renal function tests (RFTs), electrocardiogram, chest X-ray and urine analysis while thiopurine methyltransferase (TPMT) levels will be assessed specifically for group B patients. The patients will be followed up at week 4, 12 and 24. CBC, RFTs and LFTs will be done at each follow-up and EASI score will be calculated,
Period: Overall Study
Arm/Group | Methotrexate Arm | Azathioprine
Started | 10 | 10
Completed | 8 | 7
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Out of a total of 20 patients recruited, 4 were lost to follow-up (three from AZT arm and one from MTX arm). One patient developed anemia while on methotrexate and the treatment was discontinued. The final analysis included a total of 15 patients (7 from AZT arm and 8 from MTX arm).
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate Arm | Azathioprine | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants] — Population: Out of a total of 20 patients recruited, 4 were lost to follow-up (three from AZT arm and one from MTX arm). One patient developed anemia while on methotrexate and the treatment was discontinued. The final analysis included a total of 15 patients (7 from AZT arm and 8 from MTX arm).
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 4 | 3 | 7
    >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Out of a total of 20 patients recruited, 4 were lost to follow-up (three from AZT arm and one from MTX arm). One patient developed anemia while on methotrexate and the treatment was discontinued. The final analysis included a total of 15 patients (7 from AZT arm and 8 from MTX arm).
  Participants
    Female | 0 | 0 | 0
    Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
50% improvement in Eczema Area and Severity Index (EASI-50) [Mean (Full Range); unit: units on a scale] — EASI-50 implies 50% reduction in EASI score from baseline. The total EASI score is between 0 and 72 .
  Mild disease: Patients with a score of 1.1-7.0 on the EASI scale will be classified as having mild disease.
  Moderate disease: Patients with a score of 7.1 to 21.0 on the EASI scale will be classified as having moderate disease.
  Severe disease: Patients with a score of 21.1-50.0 on the EASI scale will be classified as having severe disease.
  Very Severe disease: Patients with a score of 50.1-72.0 on the EASI scale will be classified as having very severe disease. Population: Out of a total of 20 patients recruited, 4 were lost to follow-up (three from AZT arm and one from MTX arm). One patient developed anemia while on methotrexate and the treatment was discontinued. The final analysis included a total of 15 patients (7 from AZT arm and 8 from MTX arm).
  units on a scale | 25.325 [21 to 30.4] | 25.128 [14.5 to 44.7] | 25.233 [14.5 to 44.7]

OUTCOME MEASURES:

1. Primary Outcome: 50% Reduction in the Eczema Area and Severity Index Score (EASI-50)
Description: EASI-50 means 50% reduction in the Eczema Area and Severity Index score from baseline score. EASI is a scale used to evaluate the degree and severity of eczema. The total EASI score is between 0 and 72 .
  Mild disease: Patients with a score of 1.1-7.0 on the EASI scale will be classified as having mild disease.
  Moderate disease: Patients with a score of 7.1 to 21.0 on the EASI scale will be classified as having moderate disease.
  Severe disease: Patients with a score of 21.1-50.0 on the EASI scale will be classified as having severe disease.
  Very Severe disease: Patients with a score of 50.1-72.0 on the EASI scale will be classified as having very severe disease.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate Arm | Azathioprine
Number analyzed (Participants) | 8 | 7
Participants | 3 | 2

2. Secondary Outcome: Investigator Global Assessment (IGA) Score of 0-2
Description: Investigator global assessment (IGA) is a subjective measure of disease severity which is assessed by the physician on patient's visit. It ranges from 0 to 4 (0-clear, 1-almost clear, 2-mild, 3-moderate, 4-severe)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Methotrexate Arm: After the enrollment of patients and taking consent, participants will be divided in two treatment groups via lottery method. Group A will be administered oral methotrexate 10mg/week after a test dose
  Methotrexate: Methotrexate will be started at 10mg/week and
- Azathioprine: group B will be administered tablet azathioprine at a dose of 0.3mg/kg daily after. Both group of patients will be advised regarding strict sun protection measures (sunblock, hats, sunglasses etc.). The baseline investigations for both groups will include complete blood picture (CBC), liver function tests (LFTs), renal function tests (RFTs), electrocardiogram, chest X-ray and urine analysis while thiopurine methyltransferase (TPMT) levels will be assessed specifically for group B patients. The patients will be followed up at week 4, 12 and 24. CBC, RFTs and LFTs will be done at each follow-up and EASI score will be calculated,
  Azathioprine: azathioprine will be started at 0.3mg/kg. Anticipated response is after atleast 1 month so testing will be done thereafter ( after checking initial safety profile)
Arm/Group | Methotrexate Arm | Azathioprine
Number analyzed (Participants) | 8 | 7
Participants | 5 | 3

ADVERSE EVENTS:
Time Frame: From enrollment to end of followup, upto 24 weeks
Arm/Group | Methotrexate Arm | Azathioprine
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate Arm (N=10) | Azathioprine (N=10)
Anemia/pancytopenia during treatment (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Patient was withdrawn from the study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate Arm (N=10) | Azathioprine (N=10)
Body aches and myalgias (Musculoskeletal and connective tissue disorders) | 1 | 2
Gastritis, nausea, vomiting (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Lower than expected sample size may impact on the generalizability of results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT06476366/Prot_SAP_ICF_000.pdf